CLINICAL TRIAL: NCT01370655
Title: A Phase Ib, Randomized, Double-Blind, 4-Treatment, 2-Period Incomplete Block Study to Evaluate the Multiple Dose Effects of MK-7145 and Hydrochlorothiazide Compared to Placebo on Blood Pressure in Male Patients With Hypertension
Brief Title: A Study of MK-7145 Compared to Placebo and Hydrochlorothiazide for Lowering Blood Pressure in Male Participants With Hypertension (MK-7145-009)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 7145-009
Record Dates: First submitted 2011-06-08; First posted 2011-06-10 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — MK-7145; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- MK-7145 6 mg (Treatment A) (Experimental): MK-7145 3 mg (three x 1-mg MK-7145 capsules administered orally) and placebo to HCTZ (two 12.5-mg capsules) then three x 1-mg MK-7145 capsules 4 hours later, daily for 4 weeks.
  Interventions: Drug: MK-7145; Drug: Placebo to HCTZ
- MK-7145 3 mg (Treatment B) (Experimental): MK-7145 3 mg (one 2mg MK-7145 and one MK-7145 placebo capsule) then one 1-mg MK-7145 capsule and two MK-7145 placebo capsules 4 hours later and placebo to HCTZ (2 capsules once daily) daily for 4 weeks.
  Interventions: Drug: MK-7145; Drug: Placebo to MK-7145; Drug: Placebo to HCTZ
- Hydrochlorothiazide 25 mg (Treatment C) (Active Comparator): HCTZ 25 mg (two 12.5-mg capsules) and placebo to MK-7145 (one 3-mg capsule) then placebo for MK-7145 (one 3-mg capsule) 4 hours later daily for 4 weeks.
  Interventions: Drug: Hydrochlorothiazide (HCTZ); Drug: Placebo to MK-7145
- Placebo (Treatment D) (Placebo Comparator): Placebo to MK-7145 (2 x 3-mg capsules) and placebo to HCTZ 25 mg (2 capsules) then placebo to MK-7145 (2 x 3-mg capsules) 4 hours later daily for 4 weeks
  Interventions: Drug: Placebo to MK-7145; Drug: Placebo to HCTZ

INTERVENTIONS:
Drug: MK-7145
  Arms: MK-7145 3 mg (Treatment B); MK-7145 6 mg (Treatment A)
Drug: Hydrochlorothiazide (HCTZ)
  Arms: Hydrochlorothiazide 25 mg (Treatment C)
Drug: Placebo to MK-7145
  Arms: Hydrochlorothiazide 25 mg (Treatment C); MK-7145 3 mg (Treatment B); Placebo (Treatment D)
Drug: Placebo to HCTZ
  Arms: MK-7145 3 mg (Treatment B); MK-7145 6 mg (Treatment A); Placebo (Treatment D)

SUMMARY:
This study is being done to evaluate the antihypertensive efficacy and tolerability of MK-7145 in participants with mild-to-moderate hypertension.

The primary hypotheses for the study were as follows:

1. Multiple dose administration of 6-mg MK-7145 results in a reduction in systolic blood pressure (SBP) in male participants with mild to moderate hypertension that is superior to placebo, as measured by time weighted average change from baseline over 24 hours postdose (TWA0-24hrs) on dosing Day 28
2. Multiple dose administration of 6-mg MK-7145 results in a reduction in SBP in male participants with mild to moderate hypertension that is similar to hydrochlorothiazide (HCTZ), as measured by TWA0-24hrs on dosing Day 28
3. The effect of MK-7145 and HCTZ on natriuresis (UNaV) as well as SBP and diastolic blood pressure (DBP), both as measured by TWA0-24hrs, will be estimated
4. Multiple dose administration of MK-7145 for 4 weeks will be generally safe and well-tolerated.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of essential hypertension
* Body mass index (BMI) ≤35 kg/m^2
* Participant in general good health
* No history of clinically significant arrhythmias or clinically significant abnormality on electrocardiogram (ECG)
* No history of clinically significant cardiac disease
* Treatment-naïve or taking up to 2 antihypertensive therapeutic agents
* Non-smoker and/or has not used nicotine or nicotine-containing products for at least 6 months

Exclusion criteria:

* Participant has low plasma potassium
* History of stroke, chronic seizures, or major neurological disorder
* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* History of osteoporosis
* Active or history of nephrocalcinosis, nephrolithiasis or hypercalciuria
* Orthostatic change in vital sign measurements while going from a semi-recumbent to standing position accompanied by symptoms
* Functional disability that can interfere with rising from a semi-recumbent position to the standing position
* History of malignant neoplastic disease. Exceptions: (1) adequately treated non-melanomatous skin carcinoma; (2) other malignancies which have been successfully treated >10 years prior to the prestudy (screening) visit, (3) unlikely to sustain a recurrence
* Participant is unable to refrain from the use of prescription and non-prescription drugs such as high-dose aspirin (≥325 mg/day), strong/moderate Cytochrome P450 3A4 (CYP3A4) inhibitors (such as ritonavir, indinavir, nelfinavir, erythromycin, telithromycin, clarithromycin, chloramphenicol, fluconazole, ketoconazole, itraconazole, nefazodone, aprepitant, verapamil, or diltiazem) as well as strong/moderate CYP3A4 inducers (such as phenytoin, carbamazepine, oxcarbazepine, phenobarbital, efavirenz, nevirapine, etravirine, rifampicin, modafinil, St Johns Wort, cyproterone, or progestin) beginning approximately 2 weeks (or 5 half-lives), prior to administration of the initial dose of study drug until the post study visit
* Current use of non-steroidal anti-inflammatory drugs (NSAIDs) other than low dose aspirin, aluminum- or magnesium-containing antacids, sucralfate, metal cations such as iron, multivitamins containing iron or zinc that cannot be discontinued at least 2 weeks (or 5 half-lives) prior to administration of the initial dose of study drug until the post study visit
* Consumption of excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL/10 ounces], wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]) per day
* Participant consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, or other caffeinated beverages per day
* Major surgery, donation or lost 1 unit of blood (approximately 500 mL), or participation in another investigational study within 4 weeks prior to the prestudy (screening)
* History of significant multiple and/or severe allergies (including latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Regular use of any illicit drugs or history of drug abuse within approximately 6 months
* Dehydration or volume-depletion

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-06-15 (Actual); Primary Completion 2011-12-19 (Actual); Study Completion 2012-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomly assigned to 1 of 12 treatment sequences Each 4-week treatment period was separated by a wash-out of approximately 4 weeks
Groups:
- Treatment A → Treatment C: Participants received 6 mg MK-7145 for 4 weeks and then after a 4 week washout, received HCTZ 25 mg, daily, for 4 weeks
- Treatment C → Treatment A: Participants received HCTZ 25 mg daily for 4 weeks and then after a 4-week washout, received 6 mg MK-7145 daily for 4 weeks.
- Treatment A → Treatment D: Participants received 6 mg MK-7145 daily for 4 weeks and then after a 4-week washout, received Placebo MK-7145 daily for 4 weeks.
- Treatment D → Treatment A: Participants received Placebo MK-7145 daily for 4 weeks and then after a 4-week washout, received 6 mg MK-7145 daily for 4 weeks.
- Treament D → Treatment C: Participants received Placebo MK-7145 daily for 4 weeks and then after a 4-week washout, received HCTZ 25 mg placebo daily for 4 weeks.
- Treatment C → Treatment D: Participants received HCTZ 25 mg daily for 4 weeks and then after a 4-week washout, received Placebo MK-7145 daily for 4 weeks.
- Treatment A → Treatment B: Participants received 6 mg MK-7145 daily for 4 weeks and then after a 4-week washout, received 3 mg MK-7145 daily for 4 weeks.
- Treatment B → Treatment A: Participants received 3 mg MK-7145 daily for 4 weeks and then after a 4-week washout, received 6 mg MK-7145 daily for 4 weeks.
- Treatment B → Treatment C: Participants received 3 mg MK-7145 daily for 4 weeks and then after a 4-week washout, received HCTZ 25 mg daily for 4 weeks.
- Treatment C → Treatment B: Participants received HCTZ 25 mg daily for 4 weeks and then after a 4-week washout, received 3 mg MK-7145 daily for 4 weeks.
- Treatment B → Treatment D: Participants received 3 mg MK-7145 daily for 4 weeks and then after a 4-week washout, received Placebo MK-715 daily for 4 weeks.
- Treatment D → Treament B: Participants received Placebo MK-7145 daily for 4 weeks and then after a 4-week washout, received 3 mg MK-7145 daily for 4 weeks.
Period: Period 1
Arm/Group | Treatment A → Treatment C | Treatment C → Treatment A | Treatment A → Treatment D | Treatment D → Treatment A | Treament D → Treatment C | Treatment C → Treatment D | Treatment A → Treatment B | Treatment B → Treatment A | Treatment B → Treatment C | Treatment C → Treatment B | Treatment B → Treatment D | Treatment D → Treament B
Started | 7 | 7 | 3 | 3 | 3 | 4 | 4 | 4 | 3 | 2 | 3 | 3
Completed | 5 | 7 | 3 | 3 | 3 | 4 | 3 | 4 | 3 | 2 | 3 | 3
Not Completed | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Treatment A → Treatment C | Treatment C → Treatment A | Treatment A → Treatment D | Treatment D → Treatment A | Treament D → Treatment C | Treatment C → Treatment D | Treatment A → Treatment B | Treatment B → Treatment A | Treatment B → Treatment C | Treatment C → Treatment B | Treatment B → Treatment D | Treatment D → Treament B
Started | 5 | 7 | 3 | 3 | 3 | 4 | 3 | 4 | 3 | 2 | 3 | 3
Completed | 5 | 7 | 1 | 3 | 2 | 4 | 2 | 3 | 1 | 2 | 2 | 3
Not Completed | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — met protocol specified stopping criteria | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A → Treatment C | Treatment C → Treatment A | Treatment A → Treatment D | Treatment D → Treatment A | Treament D → Treatment C | Treatment C → Treatment D | Treatment A → Treatment B | Treatment B → Treatment A | Treatment B → Treatment C | Treatment C → Treatment B | Treatment B → Treatment D | Treatment D → Treament B | Total
Number analyzed (Participants) | 7 | 7 | 3 | 3 | 3 | 4 | 4 | 4 | 3 | 2 | 3 | 3 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (8.1) | 56.1 (10.9) | 58.3 (4.5) | 60.7 (3.2) | 59.3 (8.3) | 54.8 (14.7) | 60.0 (6.7) | 52.0 (9.6) | 48.3 (12.6) | 60.5 (6.4) | 50.0 (1.0) | 49.0 (9.2) | 54.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 7 | 7 | 3 | 3 | 3 | 4 | 4 | 4 | 3 | 2 | 3 | 3 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Time-weighted Average Over 24 Hours Post Dose (TWA [0-24]) in Systolic Blood Pressure (SBP)
Description: Each participant had their blood pressure monitored by continuous 24-hour ambulatory blood pressure monitoring (ABPM) on Days -1 and 28 of each treatment period. The average systolic blood pressure over the 24-hour monitoring period was calculated for baseline (Day -1) and Day 28. The difference between baseline and Day 28 was calculated and recorded.
Time Frame: Baseline and Day 28
Population: All participants who received at least 1 dose of study drug, complied with protocol sufficiently and had available data for endpoint. Participants are grouped by study drug taken at the time of the evaluation and not by randomly assigned sequence.
Measure: Least Squares Mean (90% Confidence Interval); unit: mmHg
Groups:
- MK-7145 3 mg: Participants received 3 mg MK-7145 daily for 4 weeks
- MK-7145 6 mg: Participants received 6 mg MK-7145 for 4 weeks
- HCTZ 25 mg: Participants received HCTZ 25 mg daily for 4 weeks
- Placebo: Participants received Placebo MK-7145 daily for 4 weeks
Arm/Group | MK-7145 3 mg | MK-7145 6 mg | HCTZ 25 mg | Placebo
Number analyzed (Participants) | 17 | 25 | 21 | 16
mmHg | -9.5 [-12.7 to -6.4] | -10.2 [-12.8 to -7.6] | -4.8 [-7.6 to -1.9] | -2.8 [-6.1 to 0.4]
Statistical Analysis 1: Comparison: MK-7145 6 mg vs Placebo; Type I error rate of alpha=0.10 (1-sided) is specified for testing of the hypothesis; Test type: Non-Inferiority or Equivalence — Hypothesis supported if the upper bound of the two-sided 80% confidence interval (CI; equivalent to a one-sided upper 90% CI) is ≤0 mmHg; Difference in Least square (LS) means = -7.4, 80% CI 2-sided [-10.6 to -4.1] — MK-7145 6 mg LS mean minus Placebo LS mean
Statistical Analysis 2: Comparison: MK-7145 6 mg vs HCTZ 25 mg; Type I error rate of alpha=0.05 (1-sided) is specified for testing of the hypothesis; Test type: Non-Inferiority or Equivalence — Hypothesis supported if the upper bound of the two-sided 90% CI (equivalent to a one-sided upper 95% CI) for the difference ≤ 3.8 mmHg; Difference in LS means = -5.4, 90% CI 2-sided [-9.2 to -1.6] — MK-7145 6 mg LS mean minus HCTZ 25 mg LS mean
Statistical Analysis 3: Comparison: MK-7145 3 mg vs HCTZ 25 mg; Test type: Superiority or Other; Difference in LS means = -4.8, 90% CI 2-sided [-9.0 to -0.5] — MK-7145 3 mg LS mean minus HCTZ 25 mg LS mean
Statistical Analysis 4: Comparison: MK-7145 3 mg vs Placebo; Test type: Superiority or Other; Difference in LS Means = -6.7, 90% CI 2-sided [-11.2 to -2.2] — MK-7145 3 mg LS mean minus Placebo LS mean
Statistical Analysis 5: Comparison: HCTZ 25 mg vs Placebo; Test type: Superiority or Other; Difference in LS Means = -1.9, 90% CI 2-sided [-6.2 to 2.3] — HCTZ 25 mg LS mean minus Placebo LS mean

2. Primary Outcome: Change From Baseline in Time-weighted Average Over 24 Hours Post Dose (TWA [0-24]) in Diastolic Blood Pressure (DBP)
Description: Each participant had their blood pressure monitored by continuous 24-hour ambulatory blood pressure monitoring (ABPM) on Days -1 and 28 of each treatment period. The average diastolic blood pressure over the 24-hour monitoring period was calculated for baseline (Day -1) and Day 28. The difference between baseline and Day 28 was calculated and recorded.
Time Frame: Baseline and Day 28
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: mmHg
Arm/Group | MK-7145 3 mg | MK-7145 6 mg | HCTZ 25 mg | Placebo
Number analyzed (Participants) | 17 | 25 | 21 | 16
mmHg | -4.5 [-6.7 to -2.3] | -4.3 [-6.2 to -2.5] | -1.5 [-3.5 to 0.6] | -1.1 [-3.4 to 1.2]
Statistical Analysis 1: Comparison: MK-7145 6 mg vs Placebo; Test type: Superiority or Other; Difference in LS means = -3.2, 90% CI 2-sided [-6.1 to -0.3] — MK-7145 6 mg LS mean minus Placebo LS mean
Statistical Analysis 2: Comparison: MK-7145 6 mg vs HCTZ 25 mg; Test type: Superiority or Other; Difference in LS means = -2.9, 90% CI 2-sided [-5.5 to -0.2] — MK-7145 6 mg LS mean minus HCTZ 25 mg LS mean
Statistical Analysis 3: Comparison: MK-7145 3 mg vs HCTZ 25 mg; Test type: Superiority or Other; Difference in LS means = -3.0, 90% CI 2-sided [-6.0 to -0.1] — MK-7145 3 mg LS mean minus HCTZ 25 mg LS mean
Statistical Analysis 4: Comparison: MK-7145 3 mg vs Placebo; Test type: Superiority or Other; Difference in LS means = -3.4, 90% CI 2-sided [-6.5 to -0.2] — MK-7145 3 mg LS mean minus Placebo LS mean
Statistical Analysis 5: Comparison: HCTZ 25 mg vs Placebo; Test type: Superiority or Other; Difference in LS means = -0.3, 90% CI 2-sided [-3.3 to 2.7] — HCTZ 25 mg LS mean minus Placebo LS mean

3. Primary Outcome: Change From Baseline in Urine Sodium at 24 Hours Post-dose on Day 1
Description: Urine sodium (Na) levels were measured over 24-hours on Day -1 (baseline) and on Day 1. The total amount of Na excreted in the urine for Day-1 (baseline) and Day1 were calculated and the difference between the 2 values was recorded.
Time Frame: Baseline (Day-1) and Day 1
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: mmol/day
Arm/Group | MK-7145 3 mg | MK-7145 6 mg | HCTZ 25 mg | Placebo
Number analyzed (Participants) | 17 | 25 | 21 | 16
mmol/day | 0.4 [-31.0 to 31.7] | 46.0 [20.3 to 71.7] | 64.1 [36.6 to 91.6] | -30.5 [-61.0 to -0.1]
Statistical Analysis 1: Comparison: MK-7145 6 mg vs Placebo; Type I error rate of alpha=0.10 (1-sided) is specified for testing of the hypothesis; Test type: Non-Inferiority or Equivalence — Hypothesis supported if the lower bound of the two-sided 80% CI (equivalent to a one-sided lower 90% CI) is > 89.0 mmol/day; Difference in LS means = 76.5, 80% CI 2-sided [49.2 to 103.8] — MK-7145 6 mg LS mean minus Placebo LS mean
Statistical Analysis 2: Comparison: MK-7145 3 mg vs HCTZ 25 mg; Test type: Superiority or Other; Difference in LS means = -63.7, 90% CI 2-sided [-100.8 to -26.7] — MK-7145 3 mg LS mean minus HCTZ 25 mg LS mean
Statistical Analysis 3: Comparison: MK-7145 6 mg vs HCTZ 25 mg; Test type: Superiority or Other; Difference in LS means = -18.1, 90% CI 2-sided [-49.1 to 12.9] — MK-7145 6 mg LS mean minus HCTZ 25 mg LS mean
Statistical Analysis 4: Comparison: MK-7145 3 mg vs Placebo; Test type: Superiority or Other; Difference in LS means = 30.9, 90% CI 2-sided [-7.0 to 68.7] — MK-7145 3 mg LS mean minus Placebo LS mean
Statistical Analysis 5: Comparison: HCTZ 25 mg vs Placebo; Test type: Superiority or Other; Difference in LS means = 94.6, 90% CI 2-sided [58.8 to 130.4] — HCTZ 25 mg LS mean minus Placebo LS mean

4. Primary Outcome: Percentage of Participants Who Experienced at Least 1 Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. The percentage of participants who experienced an AE during the study was summarized by study drug taken at the time of the AE.
Time Frame: Up to 14 days post last dose of each treatment period (total of 6 weeks for each treatment period)
Population: All participants who received at least 1 dose of study drug. AEs are reported by study drug taken at the time of the event and not by randomly assigned sequence.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-7145 3 mg | MK-7145 6 mg | HCTZ 25 mg | Placebo
Number analyzed (Participants) | 19 | 28 | 26 | 19
Percentage of Participants | 84.2 | 78.6 | 73.1 | 47.4

5. Primary Outcome: Percentage of Participants Who Had Study Discontinued During the Study Due to an Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. The percentage of participants who had the administration of the study drug discontinued during the study was summarized by study drug taken at the time of the AE. Participants may or may not have completed the study.
Time Frame: up to 4 weeks of each treatment period
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-7145 3 mg | MK-7145 6 mg | HCTZ 25 mg | Placebo
Number analyzed (Participants) | 19 | 28 | 26 | 19
Percentage of Participants | 0 | 10.7 | 7.7 | 5.3

6. Primary Outcome: Percentage of Participants Who Experienced at Least 1 Drug-related Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. The percentage of participants who experienced an AE that was reported as at least possibly-related to the study was summarized by study drug taken at the time of the AE.
Time Frame: Up to 14 days post last dose of each treatment period (total of 6 weeks for each treatment period)
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-7145 3 mg | MK-7145 6 mg | HCTZ 25 mg | Placebo
Number analyzed (Participants) | 19 | 28 | 26 | 19
Percentage of Participants | 52.6 | 42.9 | 42.3 | 26.3

7. Secondary Outcome: Change From Baseline in Urine Potassium at 24 Hours Post-dose on Day 28
Description: Urine potassium (K+) levels were measured over 24-hours on Day -1 and on Day 28. The total amount of K+ excreted in the urine for Day-1 (baseline) and Day 28 were calculated and the difference between the 2 values was recorded.
Time Frame: Baseline (Day -1) and Day 28
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: mmol/day
Arm/Group | MK-7145 3 mg | MK-7145 6 mg | HCTZ 25 mg | Placebo
Number analyzed (Participants) | 17 | 25 | 21 | 16
mmol/day | 0.3 [-9.2 to 9.8] | -6.5 [-14.3 to 1.3] | -2.7 [-11.3 to 6.0] | -7.6 [-17.4 to 2.2]
Statistical Analysis 1: Comparison: MK-7145 3 mg vs Placebo; Test type: Non-Inferiority or Equivalence — If the upper bound of the two-sided 80% CI (equivalent to a one-sided upper 90% CI) for the difference is <13 mmol/day the hypothesis will be supported for the 3-mg dose and testing will continue with construction of a two-sided 80% CI for the 6-mg dose (6 mg MK-7145 - placebo). The hypothesis will be supported if one or both doses meet the test criterion; Difference in LS means = 7.9, 80% CI 2-sided [-2.3 to 18.2] — MK-7145 3 mg LS mean minus Placebo LS mean
Statistical Analysis 2: Comparison: MK-7145 6 mg vs Placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 7, analysis 1]; Difference in LS means = 1.1, 80% CI 2-sided [-8.5 to 10.7] — MK-7145 6 mg LS mean minus Placebo LS mean
Statistical Analysis 3: Comparison: MK-7145 3 mg vs HCTZ 25 mg; Test type: Superiority or Other; Difference in LS means = 3.0, 90% CI 2-sided [-9.6 to 15.6] — MK-7145 3 mg LS mean minus HCTZ 25 mg LS mean
Statistical Analysis 4: Comparison: MK-7145 6 mg vs HCTZ 25 mg; Test type: Superiority or Other; Difference in LS means = -3.9, 90% CI 2-sided [-15.0 to 7.2] — MK-7145 6 mg LS mean minus HCTZ 25 mg LS mean
Statistical Analysis 5: Comparison: HCTZ 25 mg vs Placebo; Test type: Superiority or Other; Difference in LS means = 5.0, 90% CI 2-sided [-7.7 to 17.6] — HCTZ 25 mg LS mean minus Placebo LS mean

ADVERSE EVENTS:
Time Frame: up to 14 days post last dose of study drug for each treatment period
Description: All participants who received at least 1 dose of study drug. AEs are reported by study drug taken at the time of the event and not by randomly assigned sequence
Arm/Group | MK-7145 3 mg | MK-7145 6 mg | HCTZ 25 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/28 | 2/26 | 0/19
Other Adverse Events (participants affected / at risk) | 16/19 | 19/28 | 15/26 | 9/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-7145 3 mg (N=19) | MK-7145 6 mg (N=28) | HCTZ 25 mg (N=26) | Placebo (N=19)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-7145 3 mg (N=19) | MK-7145 6 mg (N=28) | HCTZ 25 mg (N=26) | Placebo (N=19)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 5 (9) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 6 (6) | 5 (5) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Blood aldosterone increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Blood uric acid increased (Investigations) | 2 (8) | 4 (15) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (5) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 5 (8) | 8 (10) | 6 (13) | 2 (3)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.